CLINICAL TRIAL: NCT04972227
Title: A Double-blinded, Randomized, Placebo-controlled, Multiple-ascending-dose Study to Assess the Safety and Pharmacokinetics of CY6463 in Participants With Stable Schizophrenia
Brief Title: Study to Assess the Safety and Pharmacokinetics of CY6463 in Participants With Stable Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tisento Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: C6463-103
Record Dates: First submitted 2021-07-15; First posted 2021-07-22 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia
Keywords: Cognitive Impairment Associated with Schizophrenia; CIAS; CY6463
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CY6463 (Experimental): CY6463 once-daily (QD) for 14 days
  Interventions: Drug: CY6463
- Placebo (Placebo Comparator): placebo QD for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CY6463 — oral tablets
  Other Names: IW-6463; Zagociguat
  Arms: CY6463
Drug: Placebo — oral tablets
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of CY6463 when administered to participants with stable schizophrenia who are on a stable antipsychotic medication regimen

ELIGIBILITY:
INCLUSION CRITERIA:

1. Provides written informed consent to participate in this study
2. Body mass index is between 18 to 40 kg/m2
3. Fluent English speaker
4. Diagnosed with schizophrenia at least 1 year ago
5. Psychiatrically stable schizophrenia with no more than moderate symptomatology
6. On a stable atypical antipsychotic regimen
7. Agrees to use effective contraception throughout the study and for at least 3 months afterward
8. Agrees to avoid using tobacco/nicotine and caffeine for several hours at a time
9. Agrees to not participate in another study of a drug or device while in this study

EXCLUSION CRITERIA:

1. Was in another study of a drug in the past 2 months
2. Fails a drug/alcohol screen, including amphetamines, barbiturates, cocaine, marijuana, methadone, methamphetamine, 3,4 methylenedioxymethamphetamine (MDMA), phencyclidine, or nonprescribed benzodiazepines or opiates
3. Has had a recent heavy smoking habit (>40 cigarettes/2 packs/day) or recently had nicotine replacement therapy
4. Has significant heart disease
5. Has hemophilia or any other bleeding/platelet dysfunction condition
6. Has hepatitis or HIV

Additional inclusion and exclusion criteria apply, per protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and TEAEs leading to study drug discontinuation | 28 (±4) days

SECONDARY OUTCOMES:
Plasma concentrations of CY6463 | up to Day 15
Pharmacokinetic (PK) parameter: area under the concentration-time curve from time zero (predose) to 24 hours postdose (AUC0-24) | up to Day 15
PK parameter: area under the concentration-time curve during a dosing interval (AUCtau) | up to Day 15
PK parameter: average concentration during a dosing interval (Cavg) | up to Day 15
PK parameter: maximum observed concentration (Cmax) | up to Day 15
PK parameter: time to maximum observed concentration (Tmax) | up to Day 15
PK parameter: minimum observed concentration (Cmin) | up to Day 15
PK parameter: apparent systemic clearance (CL/F) | up to Day 15
PK parameter: accumulation ratio based on a comparison of AUC values after single and multiple dosing (RAUC) | up to Day 15
PK parameter: accumulation ratio based on a comparison of Cmax values after single and multiple dosing (RCmax) | up to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Chickering, Study Director — Cyclerion Therapeutics
Locations (2):
- United States (2):
  - Collaborative Neuroscience Network, Long Beach, California
  - Hassman Research Institute, Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: No